CLINICAL TRIAL: NCT04171050
Title: Pudendal Enhancement of Enhanced Recovery After Surgery (ERAS) for Reconstructive Surgery (PEERS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tamara Grisales, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pudendal Enhancement of ERAS
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Pain Management
Keywords: Pain Management; Pudendal Nerve Block (PNB); Vaginal Reconstruction
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local; Anesthesia

STUDY DESIGN:
Intervention Model Description: This will be a prospective blinded randomized controlled trial. We will recruit women who are undergoing vaginal prolapse repair surgery with a Female Pelvic Medicine and Reconstructive Surgery fellowship-trained provider within the University of California, Los Angeles (UCLA) Health System.
  Women will be recruited prior to undergoing vaginal reconstructive surgery. They will then be randomized to control group with standard of care with local anesthesia used during surgery (Group 1) or PNB in addition to use of local anesthesia typically used during surgery (Group 2).
Who Masked: Participant, Care Provider
Masking Description: The providers will know what intervention the patients underwent, but the patients and the care team obtaining pain scores in the hospital will be blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Local Anesthesia (Active Comparator): Standard of care with local anesthesia used during surgery
  Interventions: Drug: Local anaesthetic
- Group 2: Local Anesthesia plus Pudendal Nerve Block (Active Comparator): Pudendal Nerve Block (PNB) in addition to local anesthesia used during surgery
  Interventions: Drug: Pudendal Nerve Block plus anesthesia

INTERVENTIONS:
Drug: Local anaesthetic — Local anesthesia injections
  Arms: Group 1: Local Anesthesia
Drug: Pudendal Nerve Block plus anesthesia — Local anesthesia injections plus a pudendal nerve block
  Arms: Group 2: Local Anesthesia plus Pudendal Nerve Block

SUMMARY:
Patients will undergo their vaginal reconstructive surgery in the usual manner, but will also be randomly assigned on the day of surgery to either receive the extra injection of numbing medication at the onset of surgery or not. The chances they will be assigned to the additional injection is 50%. Their care in the hospital and after surgery will be the same. They will participate in the study for a total of 6 weeks during which time they will be asked to complete two phone surveys, during which a provider will check in on pain level and pain medication use, and one office visit at 6 weeks. The office visit is part of their routine care and would be a scheduled visit regardless if they participated in the study or not. If they are unable to return to the office for a postoperative visit at 6 weeks, they will be contact by phone instead to obtain information on satisfaction with postoperative care, any complications after surgery, and overall how they are doing after surgery.

DETAILED DESCRIPTION:
PROTOCOL SUMMARY AND/OR SCHEMA

To determine whether administration of a PNB at time of vaginal reconstructive surgery can reduce use of narcotics and reported pain scores in the immediate postoperative period within the setting of multimodal postoperative pain control of ERAS. Women >18yo undergoing vaginal reconstructive surgery without a hysterectomy will be randomized to either standard of care with typical use of local anesthetic during their surgery versus perioperative PNB in addition to typical use of local anesthetic during their surgery. PNB will be performed with 0.5% bupivacaine and 10cc will be injected bilaterally. All patients will be on a standard preoperative and postoperative multimodal pain regimen. Patients will be followed until 6 weeks after surgery.

OVERVIEW OF STUDY DESIGN/INTERVENTION

This will be a prospective blinded randomized controlled trial. We will recruit women who are undergoing vaginal prolapse repair surgery with a Female Pelvic Medicine and Reconstructive Surgery fellowship-trained provider within the UCLA Health System. Women will be recruited prior to undergoing vaginal reconstructive surgery. They will then be randomized to control group with standard of care with local anesthesia used during surgery (Group 1) or PNB in addition to use of local anesthesia typically used during surgery (Group 2).

All pain medication will be standardized. Preoperative medications per our ERAS protocol will include oral acetaminophen 1000mg, gabapentin 600mg, and celecoxib 400mg. During surgery the patient will undergo their randomized intervention as either Group 1 or Group 2. Postoperative medications per our ERAS protocol including scheduled acetaminophen 1,000mg PO every 6 hours and ketorolac 30mg IV every 6 hours. For supplemental pain medication patients will have the following available: tramadol 50mg PO every 6 hours as needed for moderate pain (pain 4-6/10 on NRS scale), tramadol 100mg PO every 6 hours as needed for severe pain (pain 7-10/10 on NRS scale), and oxycodone 5mg PO every 4 hours as needed for breakthrough pain as supplemental pain medication. If the above regimen does not allow for sufficient pain control then additional hydromorphone IV 0.2mg or morphine IV 2mg can be ordered by the provider as needed, but will not be standard in the postoperative order set. The providers will know what intervention the patients underwent, but the patients and the care team obtaining pain scores in the hospital will be blinded to the intervention.

The patients' pain scores on the numeric rating scale (NRS) and supplemental opioid use measured in morphine milligram equivalent (MME) will be tracked during their hospitalization, which is typically a 23-hour observation. They will then be called at 48 hours for further follow-up on pain score by NRS and asked how much opioid medication they have taken since leaving the hospital and their overall satisfaction with their pain control. To help with the determination of supplemental pain medication used and pain scores, the patients will be provided a worksheet upon discharge that outlines their recommended medication routine, allows them to record their supplemental opioid medication use with dose and time, and also provides space for them to record their pain score at 48 hours post operatively. The patient will then be contacted at 2 weeks after surgery to determine if they have returned to normal activities (walking, sitting, and performing daily household tasks comfortably) and if so at what point this occurred, as well as their overall satisfaction with their postoperative pain control again. The two week contact will be either a phone call or clinic visit depending on the provider's preference for patient follow-up. The last point of contact will be at 6 weeks to determine time to return to normal activities, if they had not met this milestone at the 2-week contact, and again assess their overall satisfaction with their postoperative pain control. If a patient is discharge same day instead of admitted for 23-hour observation they will also receive a call at 24 hours postoperative to check on pain score and supplemental pain medication used.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years old
* English speaking
* Undergoing vaginal reconstructive surgery of at least 2 compartments (anterior vaginal wall, posterior vaginal wall, and/or apical suspension including hysteropexy, uterosacral ligament suspension, or sacrospinous ligament fixation)

Exclusion Criteria:

* Hysterectomy at time of surgery-is variable in duration which may affect response to PNB
* Inability to tolerate opioids-allergy or medical contraindication
* Inability to tolerate local anesthetic agents-allergy or medical contraindication
* Inability to tolerate NSAIDS-allergy or medical contraindication
* Inability to tolerate acetaminophen-allergy or medical contraindication
* Coagulation disorder
* Chronic pain syndrome using opioid medication on a regular basis prior to surgery

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women over the age of 18 undergoing vaginal reconstructive surgery without a hysterectomy
Enrollment: 44 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torosis M, Fullerton M, Kaefer D, Nitti V, Ackerman AL, Grisales T. Pudendal Block at the Time of Transvaginal Prolapse Repair: A Randomized Controlled Trial. Urogynecology (Phila). 2024 Aug 1;30(8):706-713. doi: 10.1097/SPV.0000000000001448. Epub 2024 Apr 19. PMID 38640500

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
Started | 22 | 22
Completed | 21 | 21
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Local Anesthesia: This group was assigned usual care, which involved local anesthesia administered per surgeon preference
- Total: Total of all reporting groups
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [59 to 69] | 66 [53 to 70] | 65 [58 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 16 | 34
  Black | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Other | 1 | 2 | 3
  Refused to answer | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Use
Description: Measured in morphine milligram equivalents (MME) at 24 hours
Time Frame: 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
Number analyzed (Participants) | 22 | 22
MME | 8 [0 to 20] | 6.75 [0 to 15]

2. Primary Outcome: Narcotic Use
Description: Measured in MME at 48 hours
Time Frame: 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
Number analyzed (Participants) | 22 | 22
MME | 8 [0 to 26] | 7 [0 to 35]

3. Secondary Outcome: Pain Scores
Description: Average pain score by Numerical Rating Scale (NRS). The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Time Frame: 0-2 hours, 2-4 hours, 4-8 hours, 8-12 hours, 24 hours, and 48 hours after surgery
Population: Patients were not present for 8-12 hour assessment (outpatient surgery so they were sent home)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
Number analyzed (Participants) | 22 | 22
score on a scale
  0-2 hours | 1.2 (1.8) | 1.6 (2.4)
  2-4 hours | 1.4 (1.7) | 1.1 (1.8)
  4-8 hours | 1.9 (1.8) | 1.4 (2.0)
  8-12 hours: number analyzed (Participants) | 0 | 0
  24 hours | 4 (2) | 3 (3)
  48 hours | 3 (2) | 4 (3)

4. Secondary Outcome: Return to Normal Daily Activities
Description: Days to return to normal activity, defined as walking, sitting, and performing daily household tasks comfortably. Upon discharge, all participants received a diary to record the date they returned to normal daily activities. Participants were contacted at 2 and 6 weeks postoperatively either by telephone or during their scheduled office visit and were asked about their time to return to normal activity.
Time Frame: 6 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
Number analyzed (Participants) | 22 | 22
Days | 10 [6 to 18] | 10 [7 to 11]

5. Secondary Outcome: Patient Satisfaction With Postoperative Recovery
Description: Satisfaction with postoperative pain control was assessed using a verbal scale of 1=very satisfied, 2=Somewhat satisfied, 3=Neither satisfied nor dissatisfied, 4=Somewhat dissatisfied, 5=very dissatisfied
Time Frame: 48 hours after surgery, 2 weeks after surgery
Population: Participants who completed the study, per Participant Flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
Number analyzed (Participants) | 21 | 21
Participants
  1 - at 48 hours | 16 | 13
  2 - at 48 hours | 3 | 4
  3 - at 48 hours | 0 | 1
  4 - at 48 hours | 0 | 2
  5 - at 48 hours | 1 | 0
  Not obtained at 48 hours | 1 | 1
  1 - at 2 weeks | 15 | 17
  2 - at 2 weeks | 0 | 2
  3 - at 2 weeks | 2 | 0
  4 - at 2 weeks | 0 | 1
  5 - at 2 weeks | 2 | 1
  Not obtained at 2 weeks | 2 | 0

6. Secondary Outcome: Length of Hospital Stay
Description: Tracked in hours
Time Frame: Tracked by hour through time of patient discharge (up to 72 hours)
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
Number analyzed (Participants) | 22 | 22
Hours | 16.5 [4.5 to 24] | 9 [5 to 23]

ADVERSE EVENTS:
Time Frame: 6 weeks postoperatively
Arm/Group | Group 1: Local Anesthesia | Group 2: Local Anesthesia Plus Pudendal Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/22
Other Adverse Events (participants affected / at risk) | 6/22 | 7/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Local Anesthesia (N=22) | Group 2: Local Anesthesia Plus Pudendal Nerve Block (N=22)
hospital readmission (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Local Anesthesia (N=22) | Group 2: Local Anesthesia Plus Pudendal Nerve Block (N=22)
Pudendal nerve entrapment (Surgical and medical procedures) | 0 (0) | 1 (1)
Postoperative nausea (General disorders) | 1 (1) | 0 (0)
Anesthetic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention at 48hr (Renal and urinary disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT04171050/Prot_SAP_000.pdf